CLINICAL TRIAL: NCT04802382
Title: A Phase III, Double-blind , Controlled Clinical Study Designed to Evaluate the Effect of CimetrA in Patients Diagnosed With COVID-19
Brief Title: Clinical Study Designed to Evaluate the Effect of CimetrA in Patients Diagnosed With COVID-19
Acronym: CimetrA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: MGC Pharmaceuticals d.o.o (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MGC-008
Record Dates: First submitted 2021-03-10; First posted 2021-03-17 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Corona Virus Infection; Covid19; SARS-CoV Infection
Keywords: corona; covid19; covid; coronavirus; corona virus infection; sars-cov-2
MeSH Terms: conditions — Coronavirus Infections; COVID-19; Severe Acute Respiratory Syndrome | interventions — Restraint, Physical; Hematologic Tests; Pharmacokinetics; Pregnancy Tests

STUDY DESIGN:
Intervention Model Description: Patients will be randomized in 1:1:1 ratio to one of the three arms.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 - CimetrA-1 (Experimental): a total dose containing a combination of Artemisinin 12 mg, Curcumin 40 mg, Boswellia 30 mg, and Vitamin C 120 mg in spray administration - divided into 4 separate doses given as an add on therapy, 4 doses over 48 hours (day 1 and day 2), twice a day (morning and evening).
  Interventions: Diagnostic Test: Confirm SARS-CoV-2 infection; Procedure: Physical Examination; Procedure: Vital Signs; Diagnostic Test: Hematology blood test; Diagnostic Test: Biochemistry blood test; Other: NEWS score; Diagnostic Test: PK test; Diagnostic Test: blood test for inflammatory markers; Diagnostic Test: D-dimer test; Other: VAS scale; Diagnostic Test: Urine pregnancy test for women of childbearing potential; Procedure: ECG; Other: COVID-19-Impact on Quality of Life Questionnaire; Drug: CimetrA-1
- Arm 2 - CimetrA-2 (Experimental): a total dose containing a combination of Artemisinin 8.4 mg, Curcumin 28 mg, Boswellia 21 mg, and Vitamin C 84 mg in spray administration - divided into 4 separate doses given as an add on therapy, 4 doses over 48 hours (day 1 and day 2), twice a day (morning and evening).
  Interventions: Diagnostic Test: Confirm SARS-CoV-2 infection; Procedure: Physical Examination; Procedure: Vital Signs; Diagnostic Test: Hematology blood test; Diagnostic Test: Biochemistry blood test; Other: NEWS score; Diagnostic Test: PK test; Diagnostic Test: blood test for inflammatory markers; Diagnostic Test: D-dimer test; Other: VAS scale; Diagnostic Test: Urine pregnancy test for women of childbearing potential; Procedure: ECG; Other: COVID-19-Impact on Quality of Life Questionnaire; Drug: CimetrA-2
- Arm 3 - Placebo (Placebo Comparator): composed of the same solvent but without active ingredients, given as an add on therapy in spray administration, 4 doses over 48 hours (day 1 and day 2), twice a day (morning and evening).
  Interventions: Drug: Placebo administration; Diagnostic Test: Confirm SARS-CoV-2 infection; Procedure: Physical Examination; Procedure: Vital Signs; Diagnostic Test: Hematology blood test; Diagnostic Test: Biochemistry blood test; Other: NEWS score; Diagnostic Test: PK test; Diagnostic Test: blood test for inflammatory markers; Diagnostic Test: D-dimer test; Other: VAS scale; Diagnostic Test: Urine pregnancy test for women of childbearing potential; Procedure: ECG; Other: COVID-19-Impact on Quality of Life Questionnaire

INTERVENTIONS:
Drug: Placebo administration — patients will receive the placebo treatment in addition to Standard of Care
  Arms: Arm 3 - Placebo
Diagnostic Test: Confirm SARS-CoV-2 infection — patients will be tested for SARS-CoV-2 on days 1, 14 and 28
  Other Names: Covid-19 test
Procedure: Physical Examination — patients will undergo a physical examination on days 1-14 and day 28
Procedure: Vital Signs — patient's vital signs will be measured on days 1-14 and day 28
Diagnostic Test: Hematology blood test — patients will provide a blood sample for a hematology blood test on days 1-14 and day 28
  Other Names: blood tests
Diagnostic Test: Biochemistry blood test — patients will provide a blood sample for a biochemistry blood test on days 1-14 and day 28
  Other Names: blood tests
Other: NEWS score — patient's NEWS score will be evaluated on days 1-14 and day 28
  Other Names: scoring
Diagnostic Test: PK test — PK test will be performed on day 1 only (only in Brazil sites)
  Other Names: pharmacokinetics
Diagnostic Test: blood test for inflammatory markers — patients will provide a blood sample for an inflammatory markers blood test (IL-6, IL-1β, IL-12, TNF α, IFN-γ) on days 1-7, day 14, and day 28
  Other Names: blood tests
Diagnostic Test: D-dimer test — patients will provide a blood sample for D-dimer blood test on days 1, day 2, day 7, day 14, and day 28
  Other Names: blood tests
Other: VAS scale — patient's VAS scale will be evaluated on days 1-14, day 21, and day 28
  Other Names: scoring
Diagnostic Test: Urine pregnancy test for women of childbearing potential — patients will provide a urine sample for a urine pregnancy test on days 1, and day 28
  Other Names: pregnancy test
Procedure: ECG — patients will undergo an ECG examination on days 1, and day 28
Other: COVID-19-Impact on Quality of Life Questionnaire — patients will answer the COVID-19-Impact on Quality of Life Questionnaire on days 1, 7,14,21 and 28
Drug: CimetrA-1 — patients will receive the study treatment, CimetrA-1 treatment in addition to Standard of Care
  Other Names: CimetrA-1 drug administration
  Arms: Arm 1 - CimetrA-1
Drug: CimetrA-2 — patients will receive the study treatment, CimetrA-2 treatment in addition to Standard of Care
  Other Names: CimetrA- 2 drug administration
  Arms: Arm 2 - CimetrA-2

SUMMARY:
A preparation of CimertrA, comprising Artemisinin, Curcumin, and Boswellia, and Vitamin C in a nanoparticular formulation, is proposed as a treatment for the disease associated with the novel coronavirus SARS-CoV-2. This initiative is presented under the urgent circumstances of the fulminant pandemic caused by this lethal disease, which is known as COVID-19 and has spread across the globe causing death and disrupting the normal function of modern society. The grounds for the proposal are rooted in existing knowledge on the components and pharmacological features of this formulation and their relevance to the current understanding of the disease process being addressed.

The severe acute respiratory syndrome-associated coronavirus disease 2019 (COVID-19) illness results from the immediate response to the viral infection as well as from a subsequent host inflammatory response. Systemic proinflammatory cytokines and biomarkers are elevated as the disease progresses towards its advanced stages, and correlate with worse chances of survival.

Serum cytokine levels that are elevated in patients with Covid-19-associated cytokine storm include interleukin-1β, interleukin-6, IP-10, TNF, interferon-γ, macrophage inflammatory protein (MIP) 1α and 1β, and VEGF. Higher interleukin-6 levels are strongly associated with shorter survival. The relative frequencies of circulating activated CD4+ and CD8+ T cells and plasmablasts are increased in Covid-19. In addition to the elevated systemic cytokine levels and activated immune cells, several clinical and laboratory abnormalities, such as elevated CRP and d-dimer levels, hypoalbuminemia, renal dysfunction, and effusions, are also observed in Covid-19. Laboratory test results reflecting hyper inflammation and tissue damage were found to predict worsening outcomes in Covid-19.

CimetrA, comprising Artemisinin, Curcumin, Boswellia, and Vitamin C in a nanoparticular formulation, has been studied on patients with COVID-19 in a randomized double-blind control Phase II study (MGC-006 - under a previous product name - ArtemiC). The study product demonstrated excellent safety and efficacy profiles.

Experiments performed in vitro with CimetrA demonstrated the ability to reduce cytokine elevation in response to stimulation of human PBMC preparations.

The currently proposed Multi-center multinational-controlled study is designed to include 252 adult patients who suffer from moderate COVID-19 infection. Safety will be assessed through collection and analysis of adverse events, blood and urine laboratory assessments, and vital signs.

After the screening visit, the study drug will be administrated twice a day morning and evening (every 12 hours) during (day 1 and day 2) The patients will be randomized in 1:1:1 ratio to study drug (CimetrA) in addition to Standard of Care (Arm 1 (CimetrA-1) or Arm 2 (CimetrA-2)) or Placebo in addition to Standard of Care (Arm 3).

DETAILED DESCRIPTION:
The study will take place during the patient's hospitalization due to a COVID-19 infection. The study will last up to 4 weeks, until the conclusion on day 28. In case of hospital discharge within the study period, follow-up will continue per protocol until day 28 wherever the subject will be located, performed via phone call or in-clinic, depending on the status of the patient and study schedule.

252 adult patients who suffer from COVID-19 infection and do not participate in any other clinical trial. The patient must not agree to participate in any new clinical study during the study duration. The study will take place during the patient's hospitalization due to a COVID-19 infection. The study will last up to 4 weeks, until the conclusion on day 28. In case of hospital discharge within the study period, follow-up will continue per protocol until day 28 wherever the subject will be located, performed via phone call or in-clinic, depending on the status of the patient and study schedule.

Day 1 Prior to engaging in any study procedures, the subject must meet the inclusion/exclusion criteria by history (which includes a signed declination), and review and sign an ICF. Following procedures will be performed during the visit -

* Inclusion/Exclusion criteria evaluation
* Informed Consent
* Medical History
* Concomitant Medications
* Physical Examination
* Vital Signs
* Hematology blood test (local, mandatory even if there are available results from the day before)
* Biochemistry blood test (local, mandatory even if there are available results from the day before)
* NEWS score
* PK test (brazil only, central)*
* Blood test for inflammatory markers (IL-6, IL-1β, IL-12, TNF α, IFN-γ) (local)
* D-Dimer test (local)
* VAS scale
* Urine pregnancy test for women of childbearing potential
* ECG
* COVID-19-Impact on Quality of Life Questionnaire (will be completed by the staff based on the patient answer)
* Randomization in 1:1:1 ratio to study drug (CimetrA) in addition to Standard of Care (Arm 1 (CimetrA-1) or Arm 2 (CimetrA-2)) or Placebo in addition to Standard of Care (Arm 3)
* Treatment administration (twice a day, morning and evening)
* Test for detection COVID-19 (within 5 days from admission to hospital)

Day 2

* Concomitant Medications
* AE Assessment
* Physical Examination
* Vital Signs
* Hematology blood test (local, mandatory even if there are available results from the day before)
* Biochemistry blood test (local, mandatory even if there are available results from the day before)
* NEWS score
* Blood test for inflammatory markers (IL-6, IL-1β, IL-12, TNF α, IFN-γ) (local)
* D-Dimer test (local)
* VAS scale
* Treatment administration (twice a day, morning and evening)

Days 3-6

* Concomitant Medications
* AE assessment
* Physical Examination
* Vital Signs
* Hematology blood test **
* Biochemistry blood test **
* News score **
* Blood test for inflammatory markers (IL-6, IL-1β, IL-12, TNF α, IFN-γ) (local)
* VAS scale

Day 7

* Concomitant Medications
* AE assessment
* Physical Examination
* Vital Signs
* Hematology blood test (local, mandatory even if there are available results from the day before)
* Biochemistry blood test (local, mandatory even if there are available results from the day before)
* News score
* Blood test for inflammatory markers (IL-6, IL-1β, IL-12, TNF α, IFN-γ) (local)
* D-Dimer test (local)
* VAS scale
* COVID-19-Impact on Quality of Life Questionnaire (will be completed by the staff based on the patient answer)

Days 8-13

* Concomitant Medications
* AE assessment
* Physical Examination
* Vital Signs
* Hematology blood test **
* Biochemistry blood test **
* News score **
* VAS scale

Day 14

* Concomitant Medications
* AE assessment
* Physical Examination
* Vital Signs
* Hematology blood test (local, mandatory even if there are available results from the day before)
* Biochemistry blood test (local, mandatory even if there are available results from the day before)
* News score
* Blood test for inflammatory markers (IL-6, IL-1β, IL-12, TNF α, IFN-γ) (local)
* D-Dimer test (local)
* VAS scale
* Test for detection COVID-19
* COVID-19-Impact on Quality of Life Questionnaire (will be completed by the staff based on the patient answer)

Day 21 (phone visit)

* Concomitant Medications
* AE assessment
* VAS scale
* COVID-19-Impact on Quality of Life Questionnaire (will be completed by the staff based on the patient answer)

Day 28 - Follow Up (clinic visit)

* Concomitant Medications
* AE assessment
* Physical Examination
* Vital Signs
* Hematology blood test (local, mandatory even if there are available results from the day before)
* Biochemistry blood test (local, mandatory even if there are available results from the day before)
* News score
* Blood test for inflammatory markers (IL-6, IL-1β, IL-12, TNF α, IFN-γ) (local)
* D-Dimer test (local)
* VAS scale
* Test for detection COVID-19
* Urine pregnancy test for women of childbearing potential
* ECG
* COVID-19-Impact on Quality of Life Questionnaire (will be completed by the staff based on the patient answer)

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed SARS-CoV-2 infection (according to nationally authorized laboratory criteria)
2. Hospitalized patient with COVID-19 of moderate stable or worsening severity not requiring ICU admission.
3. Age: 18 years old and above.
4. Subjects must be under observation or admitted to a controlled facility or hospital (home quarantine is not sufficient).
5. Ability to receive treatment by spray into the oral cavity

Exclusion Criteria:

1. Tube feeding or parenteral nutrition.
2. Patients with scores 5 or above per the Ordinal Scale for Clinical Improvement published by the WHO. (i.e., who need oxygen supply beyond use of nozzles or simple mask)
3. Need for admission to ICU during the present hospitalization at any time prior to completion of the recruitment to the study.
4. Any condition which, in the opinion of the Principal Investigator, would prevent full participation in this trial or would interfere with the evaluation of the trial endpoints.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2021-06-11 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
clinical improvement in treatment groups | up to 28 days
  Time to sustained clinical improvement, defined as a national Early Warning Score 2 (NEWS2) of 2 Maintained for 24 Hours in comparison to routine treatment (measured on days 7, 14, 28)

SECONDARY OUTCOMES:
oxygen dependency | up to 28 days
  Number of participants with depending on oxygen supplementation through day 28 since onset of symptoms
change in inflammatory marker levels | up to day 28
  Change in inflammatory marker levels - IL-6, IL-1β, IL-12, TNF α, IFN-γ, CRP, NLR (Neutrophil / Lymphocyte ratio) at days 1, 2, 4, 7, 14, 28
effective dose determination | up to 28 days
  Definition of the active dose of CimetrA
Pharmacokinetic profile | up to 28 days
  Pharmacokinetic profile of the study drug-AUC(mmol/L·h)
Pharmacokinetic profile | up to 28 days
  Pharmacokinetic profile of the study drug-Tmax (Hour)
Pharmacokinetic profile | up to 28 days
  Pharmacokinetic profile of the study drug-Cmax (mmol/L)
Incidence of mechanical ventilation | up to 28 days
  Incidence of mechanical ventilation
Incidence of Intensive Care Unit (ICU) stay during COVID-19 complication | up to 28 days
  Incidence of Intensive Care Unit (ICU) stay during COVID-19 complication
evaluation of drug related adverse events | up to 28 days
  Percentage of participants with definite or probable drug related adverse events
Long term adverse events of COVID-19 | up to 28 days
  Long term adverse events of COVID-19 on Day 28
Quality of life of patients | up to 28 days
  Quality of life of patients on Days 0, 14 and 28. COVID-19 - Impact on Quality of Life (COV19-QoL) scale questionnaire. The scale was made in order to serve as a tool for controlling the impact of the situation with the COVID19 pandemic in general on findings of various research on mental health.The higher score, the greater impact on quality of life and related domains subjectively perceived by the participants.
  Scores could be displayed and analyzed for each item separately. recommend the following way of calculating the total score for each participant: summing the scores on all of the items and dividing that result by the number of items (i.e. 6). Hence, the total score will be the average of all the items. The average score is measured between 1-5 scale.

OTHER OUTCOMES:
Duration of mechanical ventilation | up to day 28
  Duration of mechanical ventilation
Course of change in D Dimer levels compared to baseline | up to 28 days
Occurrence of secondary infections | up to 28 days

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Nazareth Hospital EMMS, Nazareth, North
  - Rambam Medical Center, Haifa